CLINICAL TRIAL: NCT02958917
Title: A Randomized, Double-Blind, Placebo-Controlled, Study of Efficacy and Safety of Pirfenidone in Patients With Fibrotic Hypersensitivity Pneumonitis
Brief Title: Study of Efficacy and Safety of Pirfenidone in Patients With Fibrotic Hypersensitivity Pneumonitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: covid-19 pandemic
Sponsor: Evans Fernandez Perez (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Evans Fernandez Perez, Principal Investigator, National Jewish Health
Organization: National Jewish Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-3034
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pirfenidone 2403 mg/d (Placebo Comparator): Subjects will be randomized in a 2:1 ratio to receive either pirfenidone 2403 mg/d or a placebo equivalent.
  Interventions: Drug: Pirfenidone; Other: Placebo controlled
- Placebo (Active Comparator): The placebo will be visually similar to pirfenidone.
  Interventions: Drug: Pirfenidone; Other: Placebo controlled

INTERVENTIONS:
Drug: Pirfenidone — This is a single-center, randomized, double-blind, placebo-controlled, efficacy and safety study of pirfenidone in subjects with FHP. Approximately 42-45 subjects will be randomized in a 2:1 ratio to receive pirfenidone 2403 mg/d or placebo for 52 weeks.
Other: Placebo controlled — This is a single-center, randomized, double-blind, placebo-controlled, efficacy and safety study of pirfenidone in subjects with FHP. Approximately 42-45 subjects will be randomized in a 2:1 ratio to receive pirfenidone 2403 mg/d or placebo for 52 weeks.
  Other Names: Placebo

SUMMARY:
Patients are being offered participation in this pirfenidone trial because They have been diagnosed with fibrotic hypersensitivity pneumonitis (FHP), a type of interstitial lung disease (ILD). This is a disease where scarring of lung tissue occurs as the result of inhaling substances called antigens. These antigens can be substances such as molds, chemicals or dust. As a result of this scarring the lungs are is not able to move oxygen into the bloodstream to reach other organs.

Currently over 1400 subjects have been treated with pirfenidone in 15 clinical trials. This drug has been approved by the Food and Drug Administration (FDA) for use in Idiopathic Pulmonary Fibrosis, a different type of ILD, but requires special permission for use in your condition. The use of pirfenidone has not been approved for the treatment of FHP. It is considered experimental treatment in this study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the potential benefits and the safety of treatment with pirfenidone compared to placebo in subjects with FHP.

STUDY SUMMARY This study will include about 42 subjects at National Jewish Health. This is a "double-blind study" which means neither the subject nor the study staff will know if the subject is getting pirfenidone or placebo during the study. This is done to be sure that no one knows who is getting pirfenidone or placebo and the effects of the treatment can be measured objectively, without bias. Subject's that enroll in this study will have an equal chance of getting pirfenidone or placebo. The decision about which treatment the subject will receive (randomization) is made through a central organization.

Subjects in the study will receive either pirfenidone (2403 mg every day) or placebo capsules (a safe, inactive substance that will look the same as the pirfenidone capsules). Both the placebo and pirfenidone will be supplied in opaque, hard, white gelatin capsules and will be taken as 3 capsules by mouth, 3 times a day (a total of 9 capsules per day) and should be taken with food.

Subjects who participate in this study will be asked to take the capsules as prescribed every day for 52 weeks (12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Multidisciplinary consensus diagnosis of FHP, defined from the first instance in which a patient was informed of having FHP for at least 3 to 6 months.
2. Age 18 through 80 years at randomization.
3. Diagnosis of typical or compatible FHP by HRCT according to pre-specified criteria (Note: HRCT scan performed within 6 months of the start of screening may be used if it meets image acquisition guidelines):

   a. Typical FHP: Evidence of lung fibrosis (reticular abnormality and/or, traction bronchiectasis and/or, architectural distortion, and/or honeycombing) with either of the following: i. Profuse poorly defined centrilobular nodules of ground-glass opacity affecting all lung zones.

   ii. Inspiratory mosaic attenuation with the three-density sign. AND iii. Lack of features suggesting an alternative diagnosis.

   b. Compatible FHP: Evidence of lung fibrosis (as above) with any of the following: i. Patchy or diffuse ground-glass opacity. ii. Patchy, non-profuse centrilobular nodules of ground-glass attenuation iii. Mosaic attenuation and lobular air-trapping that do not meet the criteria for typical fibrotic HP.

   AND iv. Lack of features suggesting an alternative diagnosis.

   c. Indeterminate FHP: CT signs of fibrosis without other features suggestive of HP and lack of features suggesting an alternative diagnosis. These patients are required to have a known antigen exposure and BAL lymphocytosis (≥20%) or transbronchial biopsies demonstrating non-necrotizing granuloma(s) or lymphocytosis, or surgical lung histology consistent with HP.

   FHP Disease Severity and Progression
4. FVC ≥40%, DLCO ≥30% based either on historical pulmonary function tests obtained in the 30 days prior to screening or on tests obtained during screening
5. In the investigator's opinion, evidence of disease progression: worsening respiratory symptoms and an increased in the extent of fibrosis on HRCT or relative decline in the FVC% of at least 5%.
6. Able to walk ≥100 m during the 6-minute walk test (6MWT) at Screening.

   Informed Consent and Protocol Adherence
7. Able to understand and sign a written informed consent form.
8. Able to understand the importance of adherence to study treatment and the study protocol and willing to follow all study requirements, including the concomitant medication restrictions, throughout the study

Exclusion Criteria:

* Disease-Related Exclusions

  1. Not a suitable candidate for enrollment or unlikely to comply with the requirements of this study, in the opinion of the investigator
  2. Cigarette smoking at Screening or unwilling to avoid tobacco products throughout the study
  3. Known explanation for the interstitial lung disease, including but not limited to radiation, drug toxicity, sarcoidosis, pneumoconiosis.
  4. Clinical diagnosis of any connective tissue disease, including but not limited to scleroderma, polymyositis/dermatomyositis, and rheumatoid arthritis.
  5. Expected to receive a lung transplant within 6 to12 months from randomization or on a lung transplant waiting list at randomization.

     Medical Exclusions
  6. Any condition other than FHP that, in the opinion of the investigator, is likely to result in the death of the patient within 6 to12 months.
  7. Any condition that, in the opinion of the investigator, might be significantly exacerbated by the known side effects associated with the administration of pirfenidone.
  8. Pregnancy or lactation. Women of childbearing capacity are required to have a negative serum pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using at least two methods of birth control from the date of consent through the end of the study. If abstinence is not practiced, one of the two methods of birth control should be an oral contraceptive (e.g., oral contraceptive and a spermicide).
  9. History of ongoing alcohol or substance abuse.
  10. History of severe hepatic impairment or end-stage liver disease.
  11. History of end-stage renal disease requiring dialysis.
  12. Clinical evidence of active infection including, but not limited to, bronchitis, pneumonia, sinusitis, or urinary tract infection.
  13. Unstable or deteriorating cardiac disease, including but not limited to the following:

      1. Unstable angina pectoris or myocardial infarction.
      2. Congestive heart failure requiring hospitalization.
      3. Uncontrolled clinically significant arrhythmias.

      Laboratory Exclusions
  14. Any of the following liver function test criteria above specified limits: total bilirubin > 2.0 mg/dL, excluding patients with Gilbert's syndrome; aspartate or alanine aminotransferase (AST/SGOT or ALT/SGPT) >3 ULN; alkaline phosphatase >2.5 ULN within past 30 days.
  15. Creatinine clearance <30 mL/min, calculated using the Cockcroft-Gault formula within the past 30 days.
  16. Electrocardiogram with a QTc interval >500 msec at Screening.

      Medication Exclusions
  17. Prior use of pirfenidone, nintadinib or known hypersensitivity to any of the components of study treatment.
  18. Introduction, increase or escalation of immunosuppressive pharmacological therapy within 1 month (e.g., prednisone, azathioprine, mycophenolic acid and mycophenolate mofetil).
  19. Use of any of the following therapies within 28 days before Screening:

      1. Bosentan, ambrisentan, cyclophosphamide, cyclosporine, etanercept, iloprost, infliximab, methotrexate, tacrolimus, tetrathiomolybdate, TNF-α inhibitors, imatinib mesylate, Interferon gamma-1b, and tyrosine kinase inhibitors.
      2. Fluvoxamine.
      3. Sildenafil (daily use). Note: intermittent use for erectile dysfunction is allowed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evans Fernández, MD, MS, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swigris JJ, Aronson K, Fernandez Perez ER. A first look at the reliability, validity and responsiveness of L-PF-35 dyspnea domain scores in fibrotic hypersensitivity pneumonitis. BMC Pulm Med. 2024 Apr 19;24(1):188. doi: 10.1186/s12890-024-02991-1. PMID 38641768
- [Derived] Fernandez Perez ER, Crooks JL, Lynch DA, Humphries SM, Koelsch TL, Swigris JJ, Solomon JJ, Mohning MP, Groshong SD, Fier K. Pirfenidone in fibrotic hypersensitivity pneumonitis: a double-blind, randomised clinical trial of efficacy and safety. Thorax. 2023 Nov;78(11):1097-1104. doi: 10.1136/thorax-2022-219795. Epub 2023 Apr 7. PMID 37028940
- [Derived] Fernandez Perez ER, Crooks JL, Swigris JJ, Solomon JJ, Mohning MP, Huie TJ, Koslow M, Lynch DA, Groshong SD, Fier K. Design and rationale of a randomised, double-blind trial of the efficacy and safety of pirfenidone in patients with fibrotic hypersensitivity pneumonitis. ERJ Open Res. 2021 Jun 7;7(2):00054-2021. doi: 10.1183/23120541.00054-2021. eCollection 2021 Apr. PMID 34109243

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirfenidone 2403 mg/d: Subjects will be randomized in a 2:1 ratio to receive either pirfenidone 2403 mg/d or a placebo equivalent.
  Pirfenidone: This is a single-center, randomized, double-blind, placebo-controlled, efficacy and safety study of pirfenidone in subjects with FHP. Approximately 40 subjects will be randomized in a 2:1 ratio to receive pirfenidone 2403 mg/d or placebo for 52 weeks.
  Placebo controlled: This is a single-center, randomized, double-blind, placebo-controlled, efficacy and safety study of pirfenidone in subjects with FHP. Approximately 40 subjects will be randomized in a 2:1 ratio to receive pirfenidone 2403 mg/d or placebo for 52 weeks.
- Placebo: The placebo will be visually similar to pirfenidone.
  Pirfenidone: This is a single-center, randomized, double-blind, placebo-controlled, efficacy and safety study of pirfenidone in subjects with FHP. Approximately 40 subjects will be randomized in a 2:1 ratio to receive pirfenidone 2403 mg/d or placebo for 52 weeks.
  Placebo controlled: This is a single-center, randomized, double-blind, placebo-controlled, efficacy and safety study of pirfenidone in subjects with FHP. Approximately 40 subjects will be randomized in a 2:1 ratio to receive pirfenidone 2403 mg/d or placebo for 52 weeks.
Period: Overall Study
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Started | 27 | 13
Completed (The study was terminated prematurely in December 2020 following the randomization of 40 patients due to the ongoing impacts of the COVID-19 pandemic.) | 27 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirfenidone 2403 mg/d | Placebo | Total
Number analyzed (Participants) | 27 | 13 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (6.5) | 66.5 (3.6) | 67.1 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 12 | 5 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Non-hispanic White | 25 | 12 | 37
  Hispanic/Latino | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 27 | 13 | 40
Former smoker [Number; unit: participants] | 14 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 52 in Percent Predicted FVC.
Description: The primary efficacy analysis will estimate the mean rank change in percent predicted FVC from Baseline to Week 52. Data will be analyzed using a rank linear regression model with the rank change in percent predicted FVC from Baseline to Week 52 as the outcome variable and rank Baseline percent predicted FVC and HP therapy (placebo or pirfenidone) and concomitant immunosuppressive therapy as covariates. The treatment effect will be tested using the Wald test.
  The primary efficacy analysis will be tested at an alpha level of 0.05. Missing data due to reasons other than death will be replaced with imputed values using the MICE method (multiple imputations via chained equation).
  Subjects with missing assessments due to death will be ranked worse than those who remain alive. Subjects who die will be ranked according to the time until death, with the shortest time until death as the worst rank.
Time Frame: Up to 52 weeks.
Population: The primary efficacy analysis will be analyzed using a rank linear regression model with the rank change in %FVC from Baseline to Week 52 as the outcome variable and rank Baseline %FVC and HP therapy (placebo or pirfenidone) and concomitant immunosuppressive therapy as covariates. The treatment effect will be tested using the Wald test at an alpha level of 0.05.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
percent predicted | -0.28 (8.09) | 0.58 (12.42)
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -0.76

2. Secondary Outcome: Number of Participants With Progression-free Survival (PFS) Defined as the Time From Study Treatment Randomization to the First Occurrence of Any of the Following Events:
Description: a. Relative decline from baseline in ≥10% in FVC and/or DLCO b. Acute exacerbation of FHP defined as acute respiratory declined leading to hospitalization or ER or Urgent care evaluation; or evidence of all of the following criteria within a 4-week period in the outpatient setting: i. Increase from baseline FIO2 ≥1 L O2. ii. Clinically significant worsening of dyspnea and/or cough. iii. New, superimposed ground-glass opacities or consolidation or new alveolar opacities on chest x-ray or CT.
  c. A decrease from baseline of at least 50 meters in 6mw distance. d. Change in background therapy (need for a new course of PO or IV steroids or for the patient receiving maintenance prednisone, as a need to increase the dose by 10 mg or more; and/or addition of cyclophosphamide, azathioprine, mycophenolate mofetil, or mycophenolic acid).
  e. Death
Time Frame: Up to 52 weeks.
Population: Progression-free survival was compared between the pirfenidone and placebo groups using the log-rank test. A proportional hazards model was used to estimate the hazard ratio with 95% confidence intervals.
Measure: Number; unit: participants
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
participants | 14 | 12
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Regression, Cox; Cox Proportional Hazard = 0.264

3. Secondary Outcome: Slope of FVC Over Treatment Period.
Description: The slope for the annual rate of FVC decline
Time Frame: Up to 52 weeks.
Population: The slope for the annual rate of FVC% decline will be analyzed using a random coefficient regression model with treatment and baseline FVC% as covariates
Measure: Mean (Standard Error); unit: percent predicted/year
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
percent predicted/year | 1.69 (1.57) | -0.34 (2.07)
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = 2.03

4. Secondary Outcome: Mean Change in Percent Predicted DLCO
Description: Mean change in percent predicted diffusing capacity for carbon monoxide (DLCO) from baseline to week 52
Time Frame: Up to 52 weeks.
Population: The diffusing capacity for carbon monoxide (DLCO) was analyzed using a rank linear regression model with the rank change in DLCO% predicted from baseline to week 52 as the outcome variable and rank baseline percent predicted DLCO and FHP therapy as covariates.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
percent predicted | 1.02 (12.21) | -2.12 (16.41)
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Median Difference (Final Values) = -0.108

5. Secondary Outcome: Number of Participants With All-cause Hospitalization
Description: Proportion of patients with all-cause hospitalization
Time Frame: Up to 52 weeks.
Population: logistic regression
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
Participants | 5 | 5
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Log Rank; Risk Difference (RD) = 0.364

6. Secondary Outcome: Number of Participant With Hospitalization for a Respiratory Cause
Description: The proportion of patients with hospitalization for a respiratory cause
Time Frame: Up to 52 weeks.
Population: logistic regression
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
Participants | 1 | 3
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Log Rank; Risk Difference (RD) = 0.128

7. Secondary Outcome: Visual Extent in the Percentage of Lung CT Fibrosis
Description: Mean change from baseline to week 52 in the visual extent of the percentage of lung CT fibrosis.
Time Frame: Up to 52 weeks.
Population: The visual assessment of the extent of the percentage of lung CT fibrosis will be compared between the pirfenidone and placebo groups using logistic regression accounting for possible over- or under-dispersion in the outcome. This is not a range but the percentage extent or percent amount of fibrosis visually identified by a radiologist on the lung CT.
Measure: Mean (Standard Deviation); unit: percent of fibrosis
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
percent of fibrosis | 2.22 (4.0) | 6.15 (8.45)
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -2.05

8. Other Pre Specified Outcome: St. George's Respiratory Questionnaire.
Description: Mean change from baseline in health-related quality of life, measured by SGRQ The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Time Frame: Up to 52 weeks.
Population: SGRQ baseline to 52 weeks was analyzed using a linear regression model with a separate intercept for each subject, a dichotomous time-point effect, and a multiplicative interaction between time-point and treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
score on a scale | 0.890 [-3.64 to 5.42] | 7.61 [1.08 to 14.1]
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -6.72

9. Other Pre Specified Outcome: Living With Pulmonary Fibrosis Health-Related Quality of Life
Description: Mean change from baseline in health-related quality of life, measured by the Living with pulmonary fibrosis questionnaire includes 5 subscores.
  Scores range for each of the 5 subscores go from 0 to 100, with higher scores indicating greater impairment
Time Frame: Up to 52 weeks.
Population: L-PF baseline to 52 weeks was analyzed using a linear regression model with a separate intercept for each subject, a dichotomous time-point effect, and a multiplicative interaction between time-point and treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
units on a scale
  Symptoms | 2.99 [-2.91 to 8.9] | 11.8 [3.27 to 20.3]
  Dyspnea | 1.33 [-4.63 to 7.28] | 15.6 [7.04 to 24.2]
  Energy | 2.10 [-5.60 to 9.80] | 6.28 [-4.82 to 17.4]
  Impact | -3.44 [-9.97 to 3.09] | 1.48 [-7.93 to 10.9]
  Cough | 5.56 [-3.01 to 14.1] | 5.71 [-6.64 to 18.1]
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -4.92

10. Other Pre Specified Outcome: University of California at San Diego Shortness-of-Breath Questionnaire Score.
Description: Mean change from Baseline to Week 52 in dyspnea as measured by the University of California at San Diego Shortness-of-Breath Questionnaire score.
  Scores range from 0 to 120, with higher scores indicating greater breathlessness.
Time Frame: Up to 52 weeks.
Population: UCSD-SOBQ baseline to 52 weeks was analyzed using a linear regression model with a separate intercept for each subject, a dichotomous time-point effect, and a multiplicative interaction between time-point and treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
score on a scale | 2.06 [-1.10 to 5.22] | 4.11 [-0.834 to 9.05]
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -7.92

11. Other Pre Specified Outcome: Data-driven Texture-based Quantitative Analysis of the Percent of Lung CT Fibrosis.
Description: The extent of the percentage of lung fibrosis computed by data-driven texture-based quantitative analysis. The data-driven texture-based quantitative analysis is computed as the percentage of the total lung with fibrosis.
Time Frame: Up to 52 weeks.
Population: a linear regression model with a separate intercept for each subject, a dichotomous time-point effect, and a multiplicative interaction between time-point and treatment.
Measure: Mean (95% Confidence Interval); unit: percent of fibrosis
Arm/Group | Pirfenidone 2403 mg/d | Placebo
Number analyzed (Participants) | 27 | 13
percent of fibrosis | 2.06 [-1.10 to 5.22] | 4.11 [-0.834 to 9.05]
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/d vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -2.05

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Pirfenidone 2403 mg/d | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/13
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/13
Other Adverse Events (participants affected / at risk) | 27/27 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone 2403 mg/d (N=27) | Placebo (N=13)
Nausea (Gastrointestinal disorders) | 10 | 5
Vomiting (Gastrointestinal disorders) | 5 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Gastroesophageal reflux (Gastrointestinal disorders) | 9 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Insomnia (Nervous system disorders) | 3 | 2
Fatigue (Nervous system disorders) | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Headache (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT02958917/Prot_SAP_000.pdf